CLINICAL TRIAL: NCT01657604
Title: Treatment Optimization of Newly Diagnosed Ph/BCR-ABL Positive Patients With Chronic Myeloid Leukemia (CML) in Chronic Phase With Nilotinib vs. Nilotinib Plus Interferon Alpha Induction and Nilotinib or Interferon Alpha Maintenance Therapy
Brief Title: TKI and Interferon Alpha Evaluation Initiated by the German Chronic Myeloid Leukemia Study Group - the TIGER Study
Acronym: TIGER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas Hochhaus, Chair, Dept. Hematology/Oncology, University of Jena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CML V; 2010-024262-22 (EudraCT Number)
Record Dates: First submitted 2012-07-09; First posted 2012-08-06 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML; Tasigna; Nilotinib; Interferon
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nilotinib+IFN (Experimental): Patients will receive nilotinib 300 mg BID given as two 150 mg capsules twice daily with Peginterferon α2b at a starting target dose of 30μg/week.
  Interventions: Drug: Peginterferon α2b
- Nilotinib (Active Comparator): Patients will receive nilotinib 300 mg BID given as two 150 mg capsules twice daily.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Peginterferon α2b — Patients will receive nilotinib 300 mg BID given as two 150 mg capsules twice daily with at a starting target dose of 30μg/week. After confirmed MMR or at least 24 mo. after start of therapy, maintenance therapy (nilotinib will be discontinued) will start for a study duration of up to 5 years.
  Other Names: Redipen
  Arms: Nilotinib+IFN
Drug: Nilotinib — Patients will receive nilotinib 300 mg BID given as two 150 mg capsules twice daily for a study duration of up to 5 years.
  Other Names: Tasigna
  Arms: Nilotinib

SUMMARY:
Advances in Chronic Myeloid Leukemia (CML) therapy led to an expected survival prolongation of > 20 years after diagnosis. So far, discontinuation of tyrosine kinase inhibitors led to recurrence of disease in the majority of patients. The trial aims to improve treatment strategies in CML by improving induction therapy and deescalating maintenance therapy using low dose IFN as inducer of immunosurveillance. The trial will provide important data on the duration of active therapy in CML patients. Considering the rapidly increasing prevalence of CML this is of individual but also socioeconomic importance.

DETAILED DESCRIPTION:
Objectives

Primary:

* Evaluation of the major molecular response (MMR) rate at 18 months of nilotinib compared to nilotinib+pegylated Interferon alpha (IFN) in adult patients with newly diagnosed Ph/BCR-ABL CML in chronic phase.
* Evaluation of the feasibility to discontinue drug therapy in stable deep molecular response (MR4) after nilotinib versus IFN maintenance therapy.

Secondary:

* Evaluation of the efficacy and tolerability of IFN added to nilotinib 2x300 mg/day.
* Evaluation of the efficacy and tolerability of a maintenance therapy with nilotinib versus IFN after stable MMR after at least 24 months of nilotinib therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with diagnosis of CP-CML with cytogenetic confirmation of Ph chromosome [t(9;22)(q34;q11)]
* Ph negative cases or patients with variant translocations who are BCR-ABL positive in multiplex PCR (Cross, et al 1994) are eligible as well
* ECOG performance status of < 2
* Pretreatment with hydroxyurea for 6 months and imatinib or nilotinib for a duration of up to 6 weeks is permitted
* Age ≥ 18 years old (no upper age limit given)
* Normal serum levels ≥ LLN (lower limit of normal) of potassium, magnesium, total calcium corrected for serum albumin, or corrected to within normal limits with supplements
* ASAT and ALAT ≤ 2.5 x ULN (upper limit of normal) or ≤ 5.0 x ULN if considered due to leukemia
* Alkaline phosphatase ≤ 2.5 x ULN unless considered due to leukemia
* Total bilirubin ≤ 1.5 x ULN, except known Mb. Gilbert
* Serum lipase and amylase ≤ 1.5 x ULN
* Serum creatinine ≤ 2 x ULN
* Written informed consent prior to any study procedures being performed

Exclusion Criteria:

* Known impaired cardiac function, including any of the following:

  * Left ventricular ejection fraction (LVEF) < 45%
  * Congenital long QT syndrome
  * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
* Clinically significant resting bradycardia (< 50 beats per minute)
* QTc > 450 msec on screening ECG. If QTc > 450 ms and electrolytes are not within normal ranges before nilotinib dosing, electrolytes should be corrected and then the patient rescreened for QTc criterion
* Myocardial infarction within 12 months prior to starting therapy
* Other clinical significant heart disease (e.g. unstable angina, congestive heart failure, uncontrolled hypertension)
* History of acute (i.e., within 1 year of starting study medication) or chronic pancreatitis
* Acute or chronic viral hepatitis with moderate or severe hepatic impairment (Child-Pugh scores > 6), even if controlled
* Other concurrent uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infections, acute or chronic liver and renal disease) that could cause unacceptable safety risks or compromise compliance with the protocol
* Impaired gastrointestinal function or disease that may alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting and diarrhea, malabsorption syndrome, small bowel resection or gastric by-pass surgery)
* Concomitant medications with potential QT prolongation
* Concomitant medications known to be strong inducers or inhibitors of the CYP450 isoenzyme CYP3A4
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are pregnant or breast feeding, or women of reproductive potential not employing an effective method of birth control. (Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to administration of nilotinib). Post menopausal women must be amenorrheic for at least 12 months in order to be considered of non-childbearing potential. Female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Active autoimmune disorder, including autoimmune hepatitis
* Known serious hypersensitivity reactions to peginterferon alfa-2b or interferon alfa-2b or drug excipients
* Known serious hypersensitivity reactions to nilotinib
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Patients unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 717 (Actual)
Dates: Start 2012-08-24 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
MMR rate at 18 months of nilotinib monotherapy versus nilotinib+pegylated interferon alpha | at least 18 months after start of study treatment
  rate of MMR 18 months after randomization for each study treatment
rate of continuous MMR after discontinuation of nilotinib versus pegylated interferon alpha | at least 12 months after stopping all therapy
  rate of patients with molecular relapse (loss of MMR) 12 months after discontinuation of any treatment for CML

SECONDARY OUTCOMES:
rate of CCyR and MMR | at 12, 18 and 24 months after start of treatment
Time to CCyR, MMR, MR4 and MR4.5 | date of randomization until time to endpoints or end of study duration (at least 36 months)
  this time to-event endpoints give an impression of the velocity of drug response and of the time until a certain remission should be waited for
rate of MR4 and MR4.5 during maintenance therapy and after discontinuation | start of maintenance therapy (after at least 24 months of treatment) until end of study duration (at least 36 months)
Progression-Free Survival (PFS) | at 12, 24 and 60 months after start of treatment
Rate of patients off treatment for at least 6 months | at 60 months after start of treatment
  all patients and comparison of treatment arms
safety and tolerability profile of nilotinib in comparison with nilotinib+pegylated interferon alpha and pegylated interferon alpha | time of first study treatment until 28 days after stop of study treatment (expected 36 months)
  the time of risk is the time while receiving the therapy plus 28 days thereafter
patients compliance to nilotinib based therapies | until stop of study treatment (at least 36 months)
quality of life during induction therapy with ilotinib versus nilotinib+pegylated interferon alpha and during maintenance therapy with nilotinib versus pegylated interferon alpha | during induction therapy (until at least 24 months), during maintenance therapy (until at least 36 months)
pharmacoeconomics of the treatment strategies | after end of study (expected in December 2020) (up to 8 years)
Overall Survival (OS) | at 12, 24 and 60 months after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hochhaus, Prof. MD, Principal Investigator — Jena University Hospital
Locations (112):
- University Hospital and Masaryk University Brno, Brno, Czechia
- Germany (101):
  - Universitätsklinikum Aachen Medizinische Klinik IV, Aachen
  - Gesundheitszentrum St. Marien GmbH, Onkologie/ Hämatologie Onkologisches Zentrum, Amberg
  - MVZ am Klinikum Arnsberg GmbH, Hämatologie - Internistische Onkologie, Arnsberg
  - Studienzentrum Drs. Klausmann, Aschaffenburg
  - Klinikum Augsburg, Augsburg
  - Klinikum Bayreuth GmbH, Bayreuth
  - Vivantes Netzwerk für Gesundheit GmbH, Klinikum Neukölln, Klinik für Innere Medizin - Hämatologie und Onkologie, Berlin
  - Charité CVK, CC14, Klinik für Hämatologie und Onkologie, Berlin
  - Evangelisches Klinikum Bethel, Bielefeld
  - Universitätsklinikum Bonn Med. Klinik und Poliklinik III, Hämatologie, Bonn
  - Zentrum für Ambulante Hämatologie und Onkologie, Bonn
  - Städtisches Klinikum Braunschweig gGmbh, Medizinische Klinik III - Hämatologie, Braunschweig
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - DIAKO Ev. Diakonie-Krankenhaus gGmbH, Medizinische Klinik II, Bremen
  - Klinikum Chemnitz gGmbH Klinik für Innere Medizin III, Chemnitz
  - Universitätsklinikum Köln, Cologne
  - Onkologische Schwerpunktpraxis, Dresden
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Onkologisch-Hämatologische Schwerpunktpraxis, Eisenach
  - Dr. med. Ulrich Hauch, Erfurt
  - Onkologische Schwerpunktpraxis Erlangen, Onkologie, Hämatologie, Erlangen
  - Universitätsklinikum Erlangen Medizinische Klinik 5 - Hämatologie und int. Onkologie, Erlangen
  - St.-Antonius-Hospital, Klinik für Hämatologie Onkologie, Eschweiler
  - Klinik für Hämatologie Universitätsklinikum Essen, Essen
  - Klinikum der Goethe Universität, Frankfurt
  - Universitätsklinikum Freiburg Abteilung Innere Medizin I - Hämatologie und Onkologie, Freiburg im Breisgau
  - MVZ-Osthessen GmbH Klinikum Fulda Tumorklinik, Fulda
  - Praxis Dr. med. Schmitt, Gerlingen
  - Dr. med. Hans Werner Tessen, Facharzt für Innere Medizin, Goslar
  - Georg-August Universität Göttingen Abteilung Hämatologie und Onkologie, Göttingen
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Innere, Greifswald
  - Internistische Gemeinschaftspraxis, Güstrow
  - Katholisches Krankenhaus Hagen gem. GmbH, Klinik für Hämatologie und, Hagen
  - Gemeinschaftspraxis Hämatologie und internistische, Halle
  - Universitätsklinikum Halle (Saale), Halle
  - Asklepios Klinik St. Georg, Abteilung Hämatologie, Onkologie, Stammzelltransplantation, Hamburg
  - Universitätsklinikum Hamburg- Eppendorf, Medizinische Klinik 2, Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - St. Barbara-Klinik, Standort St. Josef, Hamm
  - Mediprojekt, Gesellschaft für Medizinstatistik und Projektentwicklung, Hanover
  - Medizinische Hochschule Hannover, Klinik für Hämatologie, Hämostaseologie, Onkologie und Stammzelltransplantation, Hanover
  - Universitätsklinikum Heidelberg Innere Medizin V: Hämatologie, Onkologie und Rheumatologie, Heidelberg
  - Internistische Gemeinschaftspraxis Heilbronn, Heilbronn
  - St. Bernward Krankenhaus Hildesheim, Hildesheim
  - Universitätsklinikum des Saarlandes Klinik für Innere Medizin I, Homburg/ Saar
  - Klinikum Idar-Oberstein GmbH, Innere Medizin I (Hämatologie/Onkologie), Idar-Oberstein
  - MVZ Onkologie Ingolstadt, Ingolstadt
  - Universitätsklinikum Jena, Klinik für Innere Medizin II, Abt. Hämatologie und internistische Onkologie, Jena
  - Westpfalz-Klinikum GmbH Innere 1, Kaiserslautern
  - Städtisches Klinikum Karlsruhe gGmbH, Medizinische Klinik III: Hämatologie/Onkologie, Karlsruhe
  - St. Vincentius-Kliniken Karlsruhe, Karlsruhe
  - Klinikum Kempten Oberallgäu gGmbH, Kempten
  - Universitätsklinikum Schleswig-Holstein, II. Medizinische Klinik und Poliklinik im Städtischen Krankenhaus Kiel, Kiel
  - InVO, Institut für Versorgungsforschung in der Onkologie, Koblenz
  - Onkologische Gemeinschaftspraxis Dr. M. Neise u. Dr. A. Lollert, Krefeld
  - Onkologische Schwerpunktpraxis, Kronach
  - Onkologisches Zentrum Gemeinschaftspraxis für Hämato-/ Onkologie, Abt. für Hämato-/ Onkologie im Caritas Krankenhaus, Lebach
  - Onkologisches Schwerpunktpraxis, Leer
  - Universitätsklinikum Leipzig, Department für Innere Medizin, Leipzig
  - Dr. Aldaoud - Dr. Schwarzer Forschungsgesellschaft mbH, Leipzig
  - Krankenhausgesellschaft St. Vincenz mbH Limburg, Limburg an der Lahn
  - Gemeinschaftspraxis Uhle, Müller, Kröning, Jentsch-Ullrich, Magdeburg
  - Internistische Gemeinschaftspraxis Onkologie/Hämatologie, Mainz
  - Universitätsmedizin der Johannes- Gutenberg Universität Mainz, III. Medizinische Klinik und Poliklinik, Hämatologie, internistische Onkologie und Pneumologie, Mainz
  - Mannheimer Onkologie Praxis, Mannheim
  - Universitätsmedizin Mannheim III. Medizinische Klinik, Mannheim
  - Klinikum der Philipps-Universität Marburg, Klinik für Innere Medizin, Schwerpunkt Hämatologie, Onkologie und Immunologie, Marburg
  - Johannes Wesling Klinikum Minden, Mühlenkreikliniken (AöR), Hämatologie/Onkologie, Minden
  - Drs. Schmidt/Schauenberg Onkologie, Muhr am See
  - Stauferklinikum Schwäbisch Gmünd, Zentrum Innere Medizin, Mutlangen
  - Hämatologisch-Onkologische Gemeinschaftspraxis, München
  - Gemeinschaftspraxis Hämatologie/ Onkologie, München
  - MHP Münchener Hämatologie Praxis, München
  - Universitätsklinikum Grosshadern LMU München, München
  - Klinikum rechts der Isar, III. Medizinische Klinik und Poliklinik, München
  - Hämatologisch-Onkologische Schwerpunktpraxis, München
  - Onkologische und hämatologische Schwerpunktpraxis, Neumarkt
  - MVZ I des Klinikums Nürnberg, Nuremberg
  - Klinikum Oldenburg Klinik für Onkologie und Hämatologie / Innere Medizin II, Oldenburg
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Klinikum Passau, II. Medizinische Klinik, Passau
  - MVZ für Blut- und Krebserkrankungen, Potsdam
  - Klinikum Vest, Behandlungszentrum Recklinghausen, Medizinische Klinik III, Recklinghausen
  - Krankenhaus Barmherzige Brüder Regensburg, Klinik für Onkologie und Hämatologie, Regensburg
  - Universitätsklinikum Regensburg Abteilung für Hämatologie und internistische Onkologie, Regensburg
  - Kreiskliniken Reutlingen GmbH, Klinikum am Steinenberg, Medizinische Klinik I, Reutlingen
  - Universitätsmedizin Rostock, ZIM II Klinik für Hämatologie, Onkologie und, Rostock
  - Agaplesion Diakonieklinikum Rotenburg, Rotenburg (Wümme)
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Innere Medizin III: Sektion für Onkologie und Hämatologie, Schwäbisch Hall
  - Leopoldina-Krankenhaus, Schweinfurt
  - Klinikverbund Südwest, Kliniken Sindelfingen-Böblingen gGmbH, Sindelfingen
  - Diakonie Klinikum Stuttgart, Medizinische Klinik, Stuttgart
  - Klinikum Mutterhaus der Borromäerinnen, Trier
  - Medizinische Universitätsklinik, Department für Innere Medizin GCP Studienzentrale der Abteilung 2, Tübingen
  - Universitätsklinikum Ulm Klinik für Innere Medizin III, Ulm
  - Medizinisches Versorgungszentrum GmbH, Weiden
  - Dres. med. T. Kamp - R. Eckert Innere/Hämatologie/Onkologie, Wendlingen
  - Rems-Murr-Klinik Winnenden, Winnenden
  - Onkologische Gemeinschaftspraxis Würselen und Stolberg, Würselen
  - Universitätsklinikum Würzburg Medizinische Klinik und Poliklinik II, Würzburg
  - Heinrich-Braun-Klinikum gGmbH, Zwickau
- Switzerland (10):
  - Kantonspital Aarau AG, Aarau
  - Kantonspital Baden, Baden
  - Universitätsspital Basel, Basel
  - IOSI; Oncology Institute of Southern Switzerland, Bellinzona
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Genève, Geneva
  - Département d'oncologie UNIL-CHUV, Lausanne
  - Kantonsspital Baselland, Liestal
  - Luzerner Kantonsspital, Lucerne
  - Universitätsspital Zürich, Zurich